CLINICAL TRIAL: NCT04659460
Title: Remote Ischemic Conditioning as an Adjunct Therapy for Severe COVID-19 Disease: a Prospective Randomized Pilot Study
Brief Title: RIC as an Adjunct Therapy for Severe COVID-19 Disease: a Prospective Randomized Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Defence Research and Development Canada (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.4
Record Dates: First submitted 2020-07-03; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: COVID; Corona Virus Infection; Acute Lung Injury; Ischemia Limb; Acute Respiratory Distress Syndrome
Keywords: Remote Ischemic Conditioning; Inflammatory response
MeSH Terms: conditions — Coronavirus Infections; Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Single-centre, randomized controlled pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only Research Assistant will be unblinded. Participant, clinical team, PI, etc. will all be blinded to the randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Conditioning (Experimental): RIC interventions will be applied to the upper extremity for a total of 20 cumulative minutes of limb ischemia, at a pressure of 250 mmHg.
  Interventions: Device: Remote Ischemic Conditioning
- Sham Remote Ischemic Conditioning (Sham Comparator): RIC sham interventions will be applied to the upper extremity for a total of 20 cumulative minutes. For sham, inflation will occur.
  Interventions: Device: Remote Ischemic Conditioning

INTERVENTIONS:
Device: Remote Ischemic Conditioning — RIC interventions will be applied to the upper extremity calibrated to induce four, ten-minute cycles of five-minutes-ischemia and five-minutes-perfusion for a total of 20 cumulative minutes of limb ischemia, at a pressure of 250 mmHg.

SUMMARY:
This research aims to assess the use of an experimental and non-invasive procedure, Remote Ischemic Conditioning (RIC), as an adjunct therapy in attenuating severe COVID-19 disease. An excessive and counterproductive systemic inflammatory response is thought to be a major cause of severe disease and death in patients with COVID-19. Severe ICU cases frequently have markedly higher levels of inflammatory markers such as CRP, IL-6, IL and TNF-a; which is thought to be correlated with increasing disease severity. The relationship between dysregulated inflammatory processes and disease states such as acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) are well understood. ALI is characterized by an acute exaggerated mononuclear/neutrophilic inflammatory response followed by progressive collagen deposition in the lung, and if severe enough, may progress to ARDS requiring ventilation.

DETAILED DESCRIPTION:
This research aims to assess the use of an experimental and non-invasive procedure, Remote Ischemic Conditioning (RIC), as an adjunct therapy in attenuating severe COVID-19 disease. An excessive and counterproductive systemic inflammatory response is thought to be a major cause of severe disease and death in patients with COVID-19. Severe ICU cases frequently have markedly higher levels of inflammatory markers such as CRP, IL-6, IL-1 and TNF-a; which is thought to be correlated with increasing disease severity. The relationship between dysregulated inflammatory processes and disease states such as acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) are well understood. ALI is characterized by an acute exaggerated mononuclear/neutrophilic inflammatory response followed by progressive collagen deposition in the lung, and if severe enough, may progress to ARDS requiring ventilation.

Remote ischemic conditioning (RIC) is an experimental and non-invasive procedure that utilizes the body's natural defense against ischemia-reperfusion (IR) injury, which is believed to stimulate innate multiorgan protection against various systemic immunopathological processes. Although its mechanisms are not entirely understood, favorable outcomes have been demonstrated in multiple remote organs including the heart, kidneys, liver, and lungs. It consists of brief and repeated doses of non-lethal ischemia and reperfusion to a limb using a tourniquet, which is thought to modulate systemic inflammation by altering several inflammatory signaling pathways.

Studies have demonstrated suppression of genes encoding proteins involved in leukocyte chemotaxis, adhesion, migration, and exocytosis, as well as innate immunity responses, cytokine synthesis, and upregulation of anti-inflammatory genes. Multiple human and animal studies have demonstrated its efficacy in decreasing inflammatory biomarkers such as IL-6, CRP, IL-1B, and TNF; inflammatory mediators correlated with increasing COVID-19 disease severity. With regards to safety, currently, over 10,000 patients worldwide have completed clinical trials involving RIC, and another 20,000 are enrolled in ongoing trials. RIC presents few risks in otherwise healthy patients. Theoretical risks are highest in those patients with risk factors for vascular compromise: previous vascular surgery, vascular trauma, or known vascular disease. Excluding such patients, the practise of RIC appears to be safe in human studies This clinical trial will be enrolling 30 COVID-19+, or presumed COVID-19+ ICU patients at St. Michael's Hospital in Toronto, Canada. Eligible patients with severe COVID-19 disease will be randomized to undergo RIC versus sham-RIC. RIC interventions will be applied to one of the extremities calibrated to induce four, ten-minute cycles of five-minutes-ischemia and five-minutes-perfusion for a total of 20 cumulative minutes of limb ischemia, at a pressure of 250 mmHg. All interventions will be performed within 6 hours upon ICU admission of a confirmed or suspected COVID+ patient, given that the patient is determined eligible and their physician deems it safe to enroll. The RIC procedure will be performed every 72 hours upon randomization, +/- 1 hour to accommodate caveats in performing the procedure at that time. Blood will be collected at various timepoints to assess RIC on biomarkers of inflammation and coagulation, and clinical metrics such as need for ventilation, LOS, presentation, and timing of symptoms will be tracked. Patients not in legal capacity and when an SDM cannot be identified or contacted will be enrolled on a deferred consent basis, and provided the option of withdrawing their study data should they regain capacity.

With the current and evolving COVID-19 pandemic, ICU's are at risk of becoming overwhelmed; thus, there exists a need for a safe, rapid, and effective treatment. RIC is known to be a safe procedure that may have the potential to attenuate systemic immunopathological processes implicated in severe COVID-19 disease. If shown to be effective, it may help ameliorate the need for extensive and costly care in the ICU setting. It can theoretically be performed with any tourniquet-like device, which may be useful in a wide range of settings. Lastly, knowledge gained from this research may have the potential to inspire further work into the use of RIC in related conditions, such as viral pneumonia or sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years old
* Admission to ICU
* Either confirmed positive, or presumed, COVID-19 disease
* Radiological evidence of COVID-related pneumonia (CXR or CT abnormalities indicating COVID-19 pneumonia; such as, ground-glass opacities)
* Able to safely undergo conditioning of the arm
* No peripheral vascular disease
* No evidence of prior arm surgery
* No evidence of prior radiation or lymph node dissection
* Clinical staff deems it safe to proceed (Yes/No: signed by MRP)

Exclusion Criteria:

* Age <16 years
* Unable to safely undergo conditioning
* Known peripheral vascular disease
* Evidence of prior arm surgery
* Evidence of prior radiation or lymph node dissection
* Clinical staff deems it unsafe (Yes/No: signed by MRP)
* No radiological evidence of COVID-related pneumonia
* Hemodynamically unstable: Patients with SBP 90 or SBP 180 excluded until hemodynamically stabilized, then reassessed for inclusion
* Anti-coagulation drug use

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Interleukin 1-Beta (IL-1B) (pg/mL) | Through study completion - up to 12 months
  Serum concentration, to be collected immediately before RIC treatment, treatment plus 6 hours, treatment plus 12 hours, treatment plus 24 hours, and treatment plus 48 hours (+/- 1 hour at each 0+ time point)
Interleukin 6 (IL-6) (pg/mL) | Through study completion - up to 12 months
  Serum concentration, to be collected immediately before RIC treatment, treatment plus 6 hours, treatment plus 12 hours, treatment plus 24 hours, and treatment plus 48 hours (+/- 1 hour at each 0+ time point)
C-reactive protein (CRP) (mg/mL) | Through study completion - up to 12 months
  Serum concentration, to be collected immediately before RIC treatment, treatment plus 6 hours, treatment plus 12 hours, treatment plus 24 hours, and treatment plus 48 hours (+/- 1 hour at each 0+ time point)
Tumour Necrosis Factor Alpha (TNFa) (pg/mL) | Through study completion - up to 12 months
  Serum concentration, to be collected immediately before RIC treatment, treatment plus 6 hours, treatment plus 12 hours, treatment plus 24 hours, and treatment plus 48 hours (+/- 1 hour at each 0+ time point)
Neutrophil to Lymphocyte Ratio (NLR) (absolute neutrophils/lymphocytes) | Through study completion - up to 12 months
  Serum concentration, to be collected immediately before RIC treatment, treatment plus 6 hours, treatment plus 12 hours, treatment plus 24 hours, and treatment plus 48 hours (+/- 1 hour at each 0+ time point)
Serum Ferritin (ng/mL) | Through study completion - up to 12 months
  Serum concentration, to be collected immediately before RIC treatment, treatment plus 6 hours, treatment plus 12 hours, treatment plus 24 hours, and treatment plus 48 hours (+/- 1 hour at each 0+ time point)
International Normalized Ratio (INR) | Through study completion - up to 12 months
  Standard coagulation parameter, to be collected immediately before RIC treatment, treatment plus 6 hours, treatment plus 12 hours, treatment plus 24 hours, and treatment plus 48 hours (+/- 1 hour at each 0+ time point)
Prothrombin Time (PTT) | Through study completion - up to 12 months
  Standard coagulation parameter, to be collected immediately before RIC treatment, treatment plus 6 hours, treatment plus 12 hours, treatment plus 24 hours, and treatment plus 48 hours (+/- 1 hour at each 0+ time point)
Rotational Thromboelastometry (ROTEM) | Through study completion - up to 12 months
  ROTEM coagulation assessment using the commercial ROTEM device traditionally used for the assessment of coagulopathy, to be collected immediately before RIC treatment, treatment plus 6 hours, treatment plus 12 hours, treatment plus 24 hours, and treatment plus 48 hours (+/- 1 hour at each 0+ time point).

SECONDARY OUTCOMES:
Total duration of mechanical ventilation (number of days) | Through study completion - up to 12 months
  Number of continuous calendar days or partial calendar days including treatment with invasive ventilation.
Intensive Care Unit Length of Stay (number of days) | Through study completion - up to 12 months
  Number of continuous calendar days or partial calendar days admitted to an acute care hospital.
Hospital Length of Stay (number of days) | Through study completion - up to 12 months
  Number of continuous calendar days or partial calendar days admitted to an acute care hospital.

IPD SHARING:
Plan to Share IPD: No
Once the knowledge on RIC in severe COVID-19 patients is refined, tested, and interpreted through statistical analysis, the data will be published in a peer-reviewed journal. If deemed effective, the contextualization and adaptation may prompt a multi-center trial headed by St. Michael's Hospital to further support data. This would allow further evaluation and later implementation of the intervention with the help of the Knowledge Translation (KT) team at the Li Ka Shing Research Institute.